CLINICAL TRIAL: NCT06060080
Title: Medical Professor,CHONGQING UNIVERSITY CANCER HOSPITAL
Brief Title: Efficacy and Safety of PEG-rhG-CSF Injection for Neutrophil Reconstitution Following AHSCT in Lymphoma/Multiple Myeloma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yao Liu (Other)
Responsible Party: Sponsor-Investigator, Yao Liu, Professor, Chongqing University Cancer Hospital
Organization: Chongqing University Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023Quick review011
Record Dates: First submitted 2023-09-04; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Lymphoma; Multiple Myeloma
Keywords: PEG-rhG-CSF; Autologous Hematopoietic Stem Cell; Transplantation; Effectiveness; Safety
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical Study on PEG-rhG-CSF in the Treatment of Lymphoma/Multiple Myeloma (Experimental): In this study, lymphoma/multiple myeloma patients who meet the inclusion criteria will be administered PEG-rhG-CSF injection at a fixed dose of 6 mg on the second day after hematopoietic stem cell infusion, and the effectiveness and safety of the treatment will be observed.
  Interventions: Drug: pegylated recombinant human granulocyte-colony stimulating factor

INTERVENTIONS:
Drug: pegylated recombinant human granulocyte-colony stimulating factor — Lymphoma/multiple myeloma patients who meet the inclusion criteria will be administered PEG-rhG-CSF injection at a fixed dose of 6 mg on the second day after hematopoietic stem cell infusion, and the effectiveness and safety of the treatment will be observed.
  Other Names: PEG-rhG-CSF

SUMMARY:
This study evaluates the effectiveness and safety of PEG-rhG-CSF injection for the reconstruction of neutrophil cells after autologous hematopoietic stem cell transplantation in lymphoma/multiple myeloma patients.

DETAILED DESCRIPTION:
This study is a single-center, open-label clinical trial. Inclusion criteria involve patients with confirmed lymphoma or multiple myeloma receiving autologous hematopoietic stem cell transplantation for the first time. After calculating the sample size, an initial cohort of 40 trial patients is expected to be enrolled. Patients meeting the eligibility criteria will be assigned to receive PEG-rhG-CSF treatment on the second day after hematopoietic stem cell infusion, with a fixed dose of 6 mg. The primary outcome measure of this study is the median time for neutrophil cell reconstruction. Secondary study endpoints include safety indicators of the medication, the duration of neutrophil cell reduction (ANC≤2.0×10^9/L), the number of days patients spend in the laminar flow ward after transplantation, the usage of antibiotics, antifungal, or antiviral drugs, as well as patient expenditures, among other indicators.

Criteria for withdrawal/discontinuation of treatment:

(1) Subjects voluntarily request to withdraw from the trial;(2) Subjects who, although not explicitly requesting withdrawal from the trial, no longer adhere to the trial protocol for treatment and assessments, resulting in loss to follow-up; (3) Subjects with poor compliance who switch treatment regimens midway or use prohibited drugs within the protocol; (4) Subjects who were incorrectly enrolled; (5) Subjects experiencing intolerable allergic reactions or adverse events; (6) Subjects who pass away; (7) Other situations that meet the exclusion criteria arise.

Management of detachment cases:

When patients withdraw from the study due to allergic reactions or adverse events, researchers should take appropriate treatment measures based on the subject's condition. For mid-study withdrawal or loss to follow-up, researchers should actively take measures to complete the final assessment to analyze their efficacy and safety. All dropout cases should be documented in the case report form, and the trial conclusion form should be filled out along with the reasons for the subject dropout.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65, any gender;
2. Patients with lymphoma/multiple myeloma requiring autologous hematopoietic stem cell transplantation;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 before transplantation;
4. Basic normal function of heart, lungs, liver, and kidneys (no severe heart disease, no severe lung disease; transaminases ≤ 3× upper limit of normal, blood bilirubin ≤ 2.0 mg/dl; blood creatinine ≤ 2× upper limit of normal);
5. Pre-transplant blood counts meet the following criteria: ANC (Absolute Neutrophil Count) ≥ 1.5×10^9/L, HGB (Hemoglobin) ≥ 90g/L, PLT (Platelets) ≥ 100×10^9/L;
6. No other severe diseases that conflict with this protocol;
7. Expected survival of ≥ 3 months and willingness to follow-up;
8. Voluntary participation in this clinical trial and signing of informed consent;
9. The investigator believes that the subject will benefit from participation.

Exclusion Criteria:

1. Patients with splenomegaly;
2. Individuals who have previously undergone allogeneic or autologous hematopoietic stem cell transplantation;
3. HIV antibody-positive, HbsAg-positive, or HCV antibody-positive;
4. Impaired liver or kidney function (transaminases >3× ULN or blood bilirubin >2.0 mg/dl; blood creatinine >2× ULN);
5. Decompensated heart failure, dilated cardiomyopathy, coronary artery disease with ST-segment depression on electrocardiogram, or myocardial infarction within the last Six months;
6. Clinical symptoms of cognitive impairment or severe mental illness;
7. Allergic reactions to polyethylene glycol recombinant human granulocyte colony-stimulating factor injection or recombinant human granulocyte colony-stimulating factor injection;
8. Pregnant or breastfeeding women;
9. Investigators believe participation in this clinical trial is unsuitable.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Median time to neutrophil cell reconstruction | 0-21 days
  day-based

SECONDARY OUTCOMES:
Blood Tests | 30 days
  Counts： red blood cells [male:(4.3-5.8)×10¹²/L ),female:(3.8-5.1)×10¹²/L]; white blood cells (3.5-9.5×10^9/L); neutrophils (1.5~8.0)×10^9/L; lymphocytes (0.8-3.5)X10^9/L; and platelets (100-300)×10^9/L.
Duration of absolute neutrophil count (ANC) | 30 days
  The normal range for neutrophil count is approximately 1.8-6.3 x 10^9/L. If the ANC (Absolute Neutrophil Count) falls to ≤2.0 x 10^9/L, it is considered a possible side effect caused by the experimental drug used in this cancer patient.
Number of days staying in the laminar flow ward after transplantation | 30 days
  A laminar flow ward is used to prevent the risk of infection in patients undergoing their first autologous hematopoietic stem cell transplantation treatment.Typically, after receiving autologous hematopoietic stem cell transplantation treatment, patients reside in the Laminar flow ward for 1-3 months.
Biochemical examination | 30 days
  Alanine aminotransferase (0~40U/L), glutamine aminotransferase(<15U/L), alkaline phosphatase (40-150U/L) et al.

OTHER OUTCOMES:
Usage of antibiotics, antifungal, or antiviral medications | 100 days
  It is primarily used to prevent infections in patients' bodies following autologous hematopoietic stem cell transplantation. Record the type and dosage of medication used.
Cost | 100 days
  The total treatment cost at the time of patient discharge. Usually denominated in RMB
Incidence of adverse events | 100 days
  lack of appetite, allergic reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China